CLINICAL TRIAL: NCT07048145
Title: Effects of Pelvic Floor Muscle Exercises and Kegel Exercise Ball Utilization on Sexual Function, Urinary Incontinence and Quality of Life in Women With Pelvic Floor Muscle Weakness: A Randomized Controlled Trial
Brief Title: Effects of Kegel Ball and Pelvic Floor Exercises on Sexual Function, Unrınary Incontinence and Quality of Life in Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: sahra sultan kara (Other Government)
Responsible Party: Sponsor-Investigator, sahra sultan kara, obstetrician-gynecologist, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Organization: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Approval Number: 2024/14/889
Record Dates: First submitted 2024-12-02; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Urinary Dysfunction; Vaginal Prolapse; Sexual Function Scores; Kegel Exercises; Cystocele and Incomplete Uterovaginal Prolapse; Sexual Dysfunctions, Psychological
Keywords: pelvic floor muscle training; kegel exercise; vaginal ball; weighted ball; vaginal cones; urinary dysfuntion; sexual dysfunction
MeSH Terms: conditions — Uterine Prolapse; Cystocele; Sexual Dysfunctions, Psychological; Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two parallel groups: one receiving Kegel exercises alone and the other receiving Kegel exercises combined with the use of a vaginal Kegel ball.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kegel Exercises + Vaginal Kegel Ball (Experimental): Participants in this group will perform the same pelvic floor muscle training program as the control group, and additionally use a vaginal Kegel exercise ball during daily activities for passive pelvic stimulation.
  Interventions: Behavioral: Pelvic Floor Muscle Training
- Kegel Exercises Only (Active Comparator): Participants in this group will perform a structured 6-week pelvic floor muscle training program consisting of fast and slow contractions without the use of any device.
  Interventions: Device: Vaginal Kegel Exercise Ball

INTERVENTIONS:
Device: Vaginal Kegel Exercise Ball — A 90-gram medical-grade silicone device with internal jiggle balls used intravaginally for 30 minutes daily in the first 3 weeks and 1 hour daily in the final 3 weeks.
  Arms: Kegel Exercises Only
Behavioral: Pelvic Floor Muscle Training — Participants will perform daily Kegel exercises for 6 weeks, starting with 5 sets per day and increasing to 10 sets per day in the final 3 weeks. Each set consists of 10 fast and 10 slow contractions.
  Arms: Kegel Exercises + Vaginal Kegel Ball

SUMMARY:
Urinary incontinence and sexual dysfunction are common conditions that can significantly impact quality of life. Although surgical and medical treatments are available, many individuals seek non-invasive alternatives.

Pelvic floor muscle training, also known as Kegel exercises, aims to strengthen the pelvic muscles that support the bladder and other pelvic organs. The use of vaginal Kegel balls may enhance the effects of these exercises by promoting increased muscle activation and pelvic awareness.

Preliminary findings suggest that regular pelvic floor muscle training may improve urinary control and enhance sexual function through improved muscle strength and proprioception.

This study aims to investigate the effectiveness of pelvic floor muscle exercises and Kegel ball utilization as non-invasive options for improving pelvic health, urinary continence, and sexual well-being.

A total of 40 female participants with pelvic floor muscle weakness, urinary incontinence, and sexual dysfunction will be enrolled. All participants will undergo a physical examination. Muscle strength will be assessed using the Modified Oxford Scale, and prolapse levels, if present, will be determined using the Simplified POP-Q classification. Sociodemographic data will be collected, and participants will complete three face-to-face questionnaires.

The Sandvick Severity Index (SSI) will be used to assess the severity of urinary incontinence. The International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF), a validated questionnaire, will assess incontinence-related quality of life. The Female Sexual Function Index (FSFI), another validated instrument, will be used to assess sexual dysfunction.

Participants will be randomized by drawing from closed envelopes containing 20 cards labeled "0" and 20 labeled "1." Those who draw a "0" will be assigned to the control group and will perform pelvic floor Kegel exercises. Those who draw a "1" will be assigned to the study group, which will perform the same exercises as the control group, along with the use of a vaginal Kegel exercise ball.

All participants will receive a 6-week home-based exercise program targeting both fast-twitch (Type II) and slow-twitch (Type I) pelvic muscle fibers. The program will include fast and slow contractions, with imagery and analogies to improve comprehension. For fast contractions, the "open-close the tap" analogy will be used. For slow contractions, participants will be instructed to "squeeze while counting to five, hold for five, and relax for five," with the visualization of an elevator slowly ascending, stopping, and descending.

Each exercise set will consist of ten rapid and ten slow contractions. Participants will be instructed to perform five sets per day during the first three weeks and increase to ten sets per day in the last three weeks. This equates to a total of 50 rapid and 50 slow contractions daily in the initial phase, increasing to 100 of each by the end of the intervention.

Exercise tracking forms will be provided to allow participants to monitor compliance and document each completed session.

Participants in the study group will be given a pelvic Kegel exercise ball to use. This device is 13.5 cm in total length, with a 3.5 cm ball width, weighs approximately 90 grams, and is made of medical-grade silicone. It contains two inner jiggle balls designed to generate passive vibrations against the vaginal wall during movement, potentially stimulating pelvic muscle activity.

After receiving instruction on safe usage, participants in the study group will wear the Kegel ball for 30 minutes daily during the first three weeks, and for one hour daily during the final three weeks, while engaging in light daily activities such as walking or household movements. They will continue to perform the same exercises as the control group while integrating the device into their routine.

ELIGIBILITY:
Inclusion Criteria:

* • Women aged 18 or over

  * Suffer from stress urinary incontinence, mixed urinary incontinence, urge incontinence or urgency.
  * Being sexually active
  * Experience vaginal laxity and/or decreased sexual sensation for a period of 6 weeks or more.
  * Understand Turkish to be able to self-complete the questionnaires (validated in Turkish ).

Exclusion Criteria:

* • Not giving informed consent.

  * Has had prior surgery for incontinence, prolapse or vaginal tightening
  * Has had more than 3 urinary tract infections in the past 12 months
  * Is currently taking any medication for incontinence
  * Is pregnant or trying to become pregnant
  * Has given birth less than 6 weeks prior to enrollment
  * Has been diagnosed obese - BMI > 40
  * Has a history of neurological conditions - Parkinson's, multiple sclerosis and other
  * Women with faecal incontinence.
  * Women with grade IV prolapse.
  * Women who have perineal pain that makes it impossible to apply the spheres.
  * Not being committed to complying with a minimum of 80% of the treatment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The aim of this study is to provide an exercise-based alternative for women with pelvic floor muscle weakness, along with urinary and sexual dysfunction, by offering non-medical and non-surgical options.
  So this researh is only suitable for female gender.
Enrollment: 40 (Actual)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in Female Sexual Function Index (FSFI) Score | Baseline and 6 weeks
  Change in total FSFI score from baseline to week 6. FSFI is a validated questionnaire assessing sexual function in women, including domains of desire, arousal, lubrication, orgasm, satisfaction, and pain.
Change in International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) Score | Baseline and 6 weeks
  Change in ICIQ-SF score from baseline to week 6. ICIQ-SF assesses frequency, severity, and impact of urinary incontinence on quality of life. Higher scores indicate greater severity.
Change in Sandvick Severity Index (SSI) Score | Baseline and 6 weeks
  Change in urinary incontinence severity as measured by the Sandvick Severity Index from baseline to 6 weeks.

SECONDARY OUTCOMES:
Adherence to Exercise Program | At baseline and after 6 weeks
  Percentage of participants who completed at least 80% of the prescribed exercise sets over the 6-week period, based on self-reported tracking forms.
Feasibility and Acceptability | At baseline and after 6 weeks.
  Participant-reported acceptability of the intervention, including comfort, willingness to continue, and perceived benefit. Data collected via structured feedback form at week 6.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Healt Science, Kartal Dr. Lutfi Kirdar City Hospital, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lau HH, Su TH, Hwang JC. Impact of pelvic floor muscle training on sexual function in women affected by stress urinary incontinence. Sex Med. 2024 Jun 20;12(3):qfae040. doi: 10.1093/sexmed/qfae040. eCollection 2024 Jun. PMID 38903774
- [Background] Skaug KL, Engh ME, Bo K. Pelvic floor muscle training in female functional fitness exercisers: an assessor-blinded randomised controlled trial. Br J Sports Med. 2024 Apr 25;58(9):486-493. doi: 10.1136/bjsports-2023-107365. PMID 38413133